CLINICAL TRIAL: NCT03241875
Title: Effects of Preoperative Gabapentin Versus Pregabalin on Shoulder Pain After Laparoscopic Cholecystectomy. A Randomized Clinical Trial
Brief Title: Effects of Preoperative Gabapentin Versus Pregabalin on Shoulder Pain After Laparoscopic Cholecystectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Faculty of Medicine, Sousse (Other)
Responsible Party: Principal Investigator, Mohamed Said NAKHLI, MD, anesthesia and intensive care, Faculty of Medicine, Sousse
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Nakhli anesthesia sahloul
Record Dates: First submitted 2017-07-29; First posted 2017-08-08 (Actual); Last update posted 2017-10-02 (Actual); Status verified 2017-09

CONDITIONS: Pain, Postoperative; Cholecystectomy, Laparoscopic
Keywords: pregabalin; gabapentin; post operative pain; laparoscopic cholecystectomy
MeSH Terms: conditions — Pain, Postoperative | interventions — Pregabalin; Gabapentin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- placebo (Placebo Comparator): Patients receive 2 capsules as placebo 2 hours before anesthesia. The capsules are delivered by the hospital pharmacy.
  Interventions: Drug: Placebo oral capsule
- pregabalin (Experimental): patients receive 2 capsules of pregabalin (pregabalin 75), two hours before anesthesia.
  Interventions: Drug: Pregabalin 75mg
- gabapentin (Experimental): patients receive 2 capsules of gabapentin (gabapentin 300), two hours before anesthesia.
  Interventions: Drug: Gabapentin 300mg

INTERVENTIONS:
Drug: Pregabalin 75mg — In this group, premedication is performed with 2 capsules of pregabalin 2 hours before anesthetic induction.
  Arms: pregabalin
Drug: Gabapentin 300mg — In this group, premedication is performed with 2 capsules of gabapentin 2 hours before anesthetic induction.
  Arms: gabapentin
Drug: Placebo oral capsule — In this group, no premedication is performed, but patients receive 2 capsules of placebo 2 hours before anesthetic induction.
  Other Names: placebo
  Arms: placebo

SUMMARY:
The aim of this study is to evaluate the effect of premedication with pregabalin or gabapentin versus placebo on postoperative shoulder pain after laparoscopic cholecystectomy.

DETAILED DESCRIPTION:
Preoperative premedication with gabapentins reduces preoperative anxiety, stress response to surgical stimuli, decreases anesthetic use. The incidence of postoperative nausea and vomiting appears to be decreased. The other desired effect of gabapentins is the reduction in the intensity of postoperative pain after laparoscopic surgery.

ELIGIBILITY:
Inclusion Criteria:

* uncomplicated laparoscopic cholecystectomy
* American Society of Anesthesiologists (ASA) status < 3

Exclusion Criteria:

* acute cholecystitis
* conversion to open cholecystectomy
* history of epilepsia, psychiatric disorders and cognitive impairment
* Pregnancy and breastfeeding
* allergy to pregabalin and/or gabapentin
* Chronic pain
* Chronic medication by corticosteroids, neuroleptics or non steroidal anti inflammatory drugs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2017-08-30 (Actual); Study Completion 2017-09-28 (Actual)

PRIMARY OUTCOMES:
Post operative shoulder pain | VAS score with rest at 2h, 6h, 12h, 24h and 48 hours after surgery
  Primary outcome is the intensity of shoulder pain during the first 48 hours after laparoscopic cholecystectomy using the visual analog scale (VAS).

SECONDARY OUTCOMES:
remifentanil consumption during anesthesia | one hour after tracheal tube removal
  Remifentanil requirements during anesthesia were calculated (µg/kg/mn)
Post operative sleep quality during the first night | first night after surgery
  Patient's sleep quality was assessed during the first postoperative night by the Spiegel score.
Post operative nausea and vomiting | 2, 6, 12, 24 and 48 hours after surgery.
  The intensity of post operative nausea and vomiting was assessed by a 0 to 3 score (0: no nausea or vomiting, 1: slight mild nausea, 2: moderate nausea, 3: vomiting).

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Said Nakhli, MD, Principal Investigator — Faculty of Medicine, Sousse
Locations (1):
- Sahloul Teaching Hospital, Sousse, Tunisia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Tiippana EM, Hamunen K, Kontinen VK, Kalso E. Do surgical patients benefit from perioperative gabapentin/pregabalin? A systematic review of efficacy and safety. Anesth Analg. 2007 Jun;104(6):1545-56, table of contents. doi: 10.1213/01.ane.0000261517.27532.80. PMID 17513656
- [Result] Valadan M, Banifatemi S, Yousefshahi F. Preoperative Gabapentin to Prevent Postoperative Shoulder Pain After Laparoscopic Ovarian Cystectomy: A Randomized Clinical Trial. Anesth Pain Med. 2015 Dec 5;5(6):e31524. doi: 10.5812/aapm.31524. eCollection 2015 Dec. PMID 26705527
- [Result] Agarwal A, Gautam S, Gupta D, Agarwal S, Singh PK, Singh U. Evaluation of a single preoperative dose of pregabalin for attenuation of postoperative pain after laparoscopic cholecystectomy. Br J Anaesth. 2008 Nov;101(5):700-4. doi: 10.1093/bja/aen244. Epub 2008 Aug 20. PMID 18716003
- [Derived] Nakhli MS, Kahloul M, Jebali C, Frigui W, Naija W. Effects of Gabapentinoids Premedication on Shoulder Pain and Rehabilitation Quality after Laparoscopic Cholecystectomy: Pregabalin versus Gabapentin. Pain Res Manag. 2018 Jul 9;2018:9834059. doi: 10.1155/2018/9834059. eCollection 2018. PMID 30123399